CLINICAL TRIAL: NCT01330355
Title: Evaluation of the Safety and Efficacy of Topical Besifloxacin Ophthalmic Suspension, 0.6% Compared With Gatifloxacin, 0.3% Ophthalmic Solution for the Treatment of Presumed Bacterial Conjunctivitis in Subjects From Birth to 31 Days of Age
Brief Title: Besifloxacin Ophthalmic Suspension Verses Gatifloxacin Ophthalmic Solution in Neonates With Bacterial Conjunctivitis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 646
Record Dates: First submitted 2011-04-05; First posted 2011-04-06 (Estimated); Results first posted 2014-09-03 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-08

CONDITIONS: Bacterial Conjunctivitis
Keywords: Ocular infections, bacterial
MeSH Terms: conditions — Conjunctivitis, Bacterial; Eye Infections, Bacterial | interventions — besifloxacin; Gatifloxacin

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Besivance (Experimental): Besifloxacin 0.6% ophthalmic suspension
  Interventions: Drug: Besivance
- Gatifloxacin (Active Comparator): Gatifloxacin 0.3% ophthalmic solution
  Interventions: Drug: Gatifloxacin

INTERVENTIONS:
Drug: Besivance — Besifloxacin hydrochloride 0.6% ophthalmic suspension, one drop instilled into infected eye, three times daily (TID) for 7 days
  Arms: Besivance
Drug: Gatifloxacin — Gatifloxacin 0.3% ophthalmic solution one drop instilled into infected eye, TID for 7 days
  Arms: Gatifloxacin

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of Besivance (besifloxacin 0.6%) ophthalmic suspension compared to gatifloxacin 0.3% ophthalmic solution when administered three times daily (TID) for seven days to neonatal subjects who are 31 days or younger on the day of randomization (Visit 1).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have a clinical diagnosis of acute bacterial conjunctivitis and exhibit conjunctival discharge and redness in at least one eye. A minimum score of 1 should be present for discharge and a minimum score of 1 for conjunctival hyperemia in the same eye.

Exclusion Criteria:

* Subjects with conjunctivitis signs and/or symptoms suggestive of fungal, protozoal, or viral etiology in either eye.
* Subjects who require or are expected to require (other than study medication) use of any topical ocular medication in either eye, or systemic medications during the course of the study or prior to Day 1 specified in the protocol as ineligible.
* Subjects with any abnormality of the ocular anatomy or ocular disease/disorder specified in the protocol as ineligible.
* Subjects with systemic disease/disorder specified in the protocol as ineligible.
* Subjects who have a known or suspected poor tolerance, sensitivity, or allergy to the study medications or any of their components.
* Subjects who have a condition or are in a situation which in the investigator's opinion may impact their safety or would negatively affect the conduct or outcome of the study.

Ages: 1 Day to 31 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2011-05; Primary Completion 2013-01 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson Varughese, Study Director — Valeant/Bausch & Lomb
Locations (1):
- Bausch & Lomb Incorporated, Bridgewater, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Besivance | Gatifloxacin
Started | 16 | 17
Completed | 16 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Besivance | Gatifloxacin | Total
Number analyzed (Participants) | 16 | 17 | 33
Age, Continuous [Median (Full Range); unit: days] | 17 [6 to 26] | 14 [5 to 25] | 14 [5 to 26]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 7 | 19
  Male | 4 | 10 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 12 | 12 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Clinical Resolution
Description: Clinical resolution defined as the absence of both conjunctival discharge and conjunctival hyperemia.
Time Frame: Visit 5 (Day 8+1)
Population: The analysis population only includes those for whom the outcome was measured within the specified time frame.
Measure: Number; unit: participants
Arm/Group | Besivance | Gatifloxacin
Number analyzed (Participants) | 16 | 16
participants | 12 | 12

2. Secondary Outcome: Clinical Resolution
Description: Clinical resolution defined as the absence of both conjunctival discharge and conjunctival hyperemia.
Time Frame: Visit 3 (Day 3)
Population: The analysis population only includes those for whom the outcome was measured within the specified time frame.
Measure: Number; unit: participants
Arm/Group | Besivance | Gatifloxacin
Number analyzed (Participants) | 16 | 16
participants | 3 | 5

3. Secondary Outcome: Microbial Eradication
Description: Eradication defined as the absence of all accepted ocular bacterial species (as measured on the ordinal scale) that were present at or above threshold at baseline
Time Frame: Visit 5 (Day 8+1)
Population: The analysis population only includes those for whom the outcome was measured within the specified time frame.
Measure: Number; unit: participants
Arm/Group | Besivance | Gatifloxacin
Number analyzed (Participants) | 13 | 9
participants | 12 | 8

4. Secondary Outcome: Microbial Outcome
Description: Microbial outcome for the following groups of accepted ocular bacterial species that were present at or above threshold at baseline:
  * over all bacterial species
  * over all and individual gram-positive bacterial species
  * over all and individual gram-negative bacterial species
Time Frame: Visit 3 (Day 3) and Visit 5 (Day 8+1)
Population: The analysis population only includes those for whom the outcome was measured within the specified time frame. A subject may have tested positive for multiple bacterial species (up to 5 species).
Measure: Number; unit: events
Arm/Group | Besivance | Gatifloxacin
Number analyzed (Participants) | 13 | 9
events
  Visit 3 (Day 3) Gram-Positive | 16 | 6
  Visit 3 (Day 3) Gram-Negative | 6 | 3
  Visit 5 (Day 8) Gram-Positive | 17 | 12
  Visit 5 (Day8) Gram-Negative | 6 | 4

ADVERSE EVENTS:
Time Frame: The period of observation for collection of AEs extended from the time the subject's parent/legally authorized representative provided informed consent until the last study visit, Visit 5.
Arm/Group | Besivance | Gatifloxacin
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/17
Other Adverse Events (participants affected / at risk) | 0/16 | 5/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Besivance (N=16) | Gatifloxacin (N=17)
Conjunctivitis Bacterial (Eye disorders) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Irritability (Psychiatric disorders) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acne Infantile (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For a period of ten years, the PI agrees to keep confidential and not disclose, without the prior written consent of Sponsor, to any third party or use any technology, data, reports, results of clinical studies conducted under this Study or other information received by Sponsor, or any technology, data, reports, study materials, or other information developed by Sponsor unless disclosure by PI is required by law.